CLINICAL TRIAL: NCT03407612
Title: The Effect of Continuous Passive Motion on Pain Control Following Hip Arthroscopy
Brief Title: Outcomes of CPM Usage Following Arthroscopic Acetabular Labral Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, John Ryan, Medical Doctor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011H0416
Record Dates: First submitted 2018-01-09; First posted 2018-01-23 (Actual); Results first posted 2018-08-02 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Femoro Acetabular Impingement; Pain, Postoperative; Hip Labral Tear
Keywords: continuous passive motion device; HOS-ADL; hip arthroscopy
MeSH Terms: conditions — Femoracetabular Impingement; Pain, Postoperative | interventions — Motion Therapy, Continuous Passive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CPM (Active Comparator): These subjects received a continuous passive motion (CPM) device and were instructed to use it for 4-6 hours daily throughout the first two postoperative weeks following their arthroscopic labral repair. They were provided adequate education on how to operate the device. The subjects recorded their average usage of the CPM, as well as their personal perception of the CPM, at the postoperative 2 day, 7 day, and 14 day marks.
  Interventions: Device: Continuous Passive Motion
- No CPM (No Intervention): No CPM was administered to these subjects.

INTERVENTIONS:
Device: Continuous Passive Motion — CPM devices are used in postoperative rehabilitation and are throughout to reduce joint stiffness.
  Arms: CPM

SUMMARY:
The purpose of this study is to measure whether CPM (continuous passive motion) usage improves outcomes following arthroscopic hip surgery that includes labral repair. Investigators tested the hypothesis that CPM usage reduces pain levels and pain medication use and improves function in individuals who undergo hip arthroscopy.

DETAILED DESCRIPTION:
Subjects undergoing primary hip arthroscopy for acetabular labral repair were randomized to determine whether they would receive a CPM. Those subjects receiving a CPM were instructed to use it for 4-6 hours daily throughout the first two postoperative weeks. The total number of pain medications and average pain scores over the two weeks, as well as Hip Outcome Score Activity of Daily Living (HOS ADL) scores at standard time points were compared via a two sample t-test and intention-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* undergoing hip arthroscopy to repair a torn labrum

Exclusion Criteria:

* pregnancy
* revision surgery
* bilateral surgery

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2013-02-15 (Actual); Primary Completion 2015-06-25 (Actual); Study Completion 2015-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Ryan, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CPM Used: These subjects received a continuous passive motion (CPM) device and were instructed to use it for 4-6 hours daily throughout the first two postoperative weeks following their arthroscopic labral repair. They were provided adequate education on how to operate the device. The subjects recorded their average usage of the CPM, as well as their personal perception of the CPM, at the postoperative 2 day, 7 day, and 14 day marks.
  Continuous Passive Motion: CPM devices are used in postoperative rehabilitation and are throughout to reduce joint stiffness.
- No CPM Used: No CPM was administered to these subjects.
Period: Overall Study
Arm/Group | CPM Used | No CPM Used
Started | 19 | 23
Completed | 19 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CPM Used | No CPM Used | Total
Number analyzed (Participants) | 19 | 23 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (10.7) | 29.5 (11.1) | 32.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 1 | 3 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 19 | 23 | 42
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.5 (7.0) | 25.1 (4.6) | 26.2 (5.8)
Hand Dominance [Count of Participants; unit: Participants]
  Right Handed | 11 | 13 | 24
  Left Handed | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient Satisfaction and Functional Outcome
Description: Hip Outcome Score Activities of Daily Living (HOS ADL) questionnaire completed at specific time points. Completion of the HOS ADL provides a score from 0 to 100, with a higher score corresponding to greater level of function. The improvement preoperative to 6 month postoperative scores was also computed.
Time Frame: Baseline and 6 weeks, 12 weeks, and 6 months postoperatively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CPM Used | No CPM Used
Number analyzed (Participants) | 19 | 23
units on a scale
  Preoperative | 64.5 (11.6) | 62.7 (15.0)
  6 weeks postoperative | 74.6 (14.8) | 72.8 (12.5)
  12 weeks postoperative | 81.1 (14.6) | 81.5 (11.4)
  6 months postoperative | 81.9 (16.4) | 82.8 (12.8)
  Improvement | 17.0 (16.0) | 20.2 (15.3)
Statistical Analysis 1: Comparison: CPM Used vs No CPM Used; This analysis considers the baseline HOS-ADL measures; Test type: Equivalence — p < 0.05 required for groups to have non-equivalent results; p = 0.67, t-test, 2 sided
Statistical Analysis 2: Comparison: CPM Used vs No CPM Used; This analysis considers the 6 week postoperative HOS-ADL measures; Test type: Equivalence — p < 0.05 required for groups to have non-equivalent results; p = 0.73, t-test, 2 sided
Statistical Analysis 3: Comparison: CPM Used vs No CPM Used; This analysis considers the 12 week postoperative HOS-ADL measures; Test type: Equivalence — p < 0.05 required for groups to have non-equivalent results; p = 0.87, t-test, 2 sided
Statistical Analysis 4: Comparison: CPM Used vs No CPM Used; This analysis considers the 6 month postoperative HOS-ADL measures; Test type: Equivalence — p < 0.05 required for groups to have non-equivalent results; p = 0.78, t-test, 2 sided

2. Secondary Outcome: Analgesic Usage
Description: Analgesic usage measured via the morphine-equivalent dose of consumed analgesic medications
Time Frame: Initial two postoperative weeks
Measure: Mean (Standard Deviation); unit: morphine equivalent doses
Arm/Group | CPM Used | No CPM Used
Number analyzed (Participants) | 19 | 23
morphine equivalent doses | 239 (269) | 330 (227)
Statistical Analysis 1: Comparison: CPM Used vs No CPM Used; Test type: Equivalence — p < 0.05 required for groups to have non-equivalent results; p = 0.25, t-test, 2 sided

3. Secondary Outcome: Pain Level
Description: Change in pain level measured on a Likert-type scale from 0 to 10, with higher scores representing higher pain levels.
Time Frame: Initial two postoperative weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CPM Used | No CPM Used
Number analyzed (Participants) | 19 | 23
units on a scale | 2.94 (2.0) | 4.23 (2.0)
Statistical Analysis 1: Comparison: CPM Used vs No CPM Used; Test type: Equivalence — p < 0.05 required for groups to have non-equivalent results; p = 0.04, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months from operation date
Arm/Group | CPM Used | No CPM Used
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/23
Other Adverse Events (participants affected / at risk) | 0/19 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes